CLINICAL TRIAL: NCT05281809
Title: A Feasibility Study Following a Phase 2a Design to Demonstrate Successful Local Manufacture of Chimeric Antigen Receptor (CAR) T-Cell Products for the Treatment of B-Cell Lymphoma and B-Acute Lymphoblastic Leukemia
Brief Title: Local Manufacture of CAR T-Cell Products for the Treatment of B-Cell Lymphoma and B-Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John Lister (Other)
Collaborators: Lentigen Technology, Inc. (Unknown); Miltenyi Biotec, Inc. (Industry); Allegheny Health Network (Other)
Responsible Party: Sponsor-Investigator, John Lister, Chief, Division of Hematology and Cellular Therapy at Allegheny Health Network, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Organization: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-114-WPH
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: B-Cell Lymphoma; B Acute Lymphoblastic Leukemia; Diffuse Large B Cell Lymphoma; Mantle Cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Lymphoplasmacytic Lymphoma; Chronic Lymphocytic Leukemia; Transformed Lymphoma
Keywords: CAR T-cell; CD19 (cluster of differentiation antigen) 19
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Receptors, Chimeric Antigen; Automobiles

STUDY DESIGN:
Intervention Model Description: administration of locally manufactured cd19-targeted CAR T-cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): CAR -T-cell collection, infusion
  Interventions: Drug: Chimeric Antigen Receptor (CAR) T-Cell Product (Autologous)

INTERVENTIONS:
Drug: Chimeric Antigen Receptor (CAR) T-Cell Product (Autologous) — This protocol describes the use of an automated cell processor and culture system, the CliniMACS Prodigy device sold by Miltenyi Biotec, for the local manufacture of CAR T-cells targeting the CD19 antigen. The manufacturing process will use a lentiviral vector (CAR19) provided by Lentigen, a wholly owned subsidiary of Miltenyi Biotec, to transfect T-cells collected from eligible patients. Live cells will be harvested by the device after culture and infused intravenously to the patient from whom the cells were originally obtained.

SUMMARY:
This trial aims to demonstrate the feasibility of this approach to reliably generate product and to safely administer the product to patients who have B-Cell Lymphoma and B-Acute Lymphoblastic Leukemia.

DETAILED DESCRIPTION:
On this study the following procedures are sequentially performed: eligibility determination and informed consent; cell collection by apheresis; CAR T-cell manufacturing and lymphodepleting chemotherapy all followed by CAR T-cell infusion on day 0. The first 3 subjects will be followed in hospital from day 0 until +14 for CRS, ICANS and other toxicity. The PI and two physicians not affiliated with the study (Nathan Bahary, MD, PhD and Gene Finley, MD) will review the outcome of the first three patients to assure the interim analysis meets criteria for continuing accrual. This analysis will be submitted to the IRB prior to continuing with accrual. The toxicity profile of the first three subjects will be scrutinized. Should toxicity be minimal with CRS ≤ 2 and ICANS grade ≤1 then the PI might propose modification to hospitalization between days 0 and +14 according to comparison with prior experience with commercially available product. A protocol amendment would be submitted in this case. Should no CAR T-cell related toxicity be identified on day +15, the subject will be discharged from the hospital and followed in the Medical Short Stay Unit (or designated substitute inpatient unit) daily to day 30. At the discretion of the Investigator (based upon each subject's medical condition or status), this follow-up could be reduced to thrice weekly basis (e.g. Monday-Wednesday-Friday). CAR T-cell monitoring by flow cytometry will occur on day +30 and day +100. Response will be assessed at day +30 and the subject will be discharged for outpatient follow up. Response will be assessed monthly by clinical examination to day +100 and then every 3 months to day +730. Thereafter, clinical follow up will occur every 6 months to five years and then yearly up to 15 years, or until death (whichever occurs first). All subjects treated on this study must consent to reporting of de-identified data to the Center for International Blood and Marrow Transplantation Research (CIBMTR). (See Table 1: Schedule of Study Procedures, Figure 1: Study Diagram, Table 2: Laboratory Investigation and Table 3: Response Evaluation for details of study conduct.) The clinical care of subjects enrolled on this study is entirely within the standard of care employed for patients who receive commercial product. There are no drugs, surgical procedures, radiological investigations, laboratory tests or examinations that are considered experimental except for a peripheral blood sample to detect CAR T-cells (by flow cytometry) and the actual production/manufacture of CAR T-cells occurring in the local Cell Processing Laboratory.

For this reason, the intent of this protocol is to ensure that the standard of care is strictly followed as outlined in the SOP documents, screenshots and documents included in the appendix of this document. Thus, patients receiving commercial product and those treated on this protocol should receive the same supportive care. In addition to immune effector cells, these documents often describe methods and cellular therapy products not relevant to this investigation and for our purpose these sections can be ignored.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with CD19+ B-cell lymphoma or B-Cell Acute Lymphoblastic Leukemia (B-ALL) with no currently available curative treatment option (such as autologous or allogeneic Hematopoietic stem cell transplantation (HSCT)) who have a limited prognosis (<2-year projected survival) will be enrolled. Participation on this trial is permitted as a bridge to HSCT.
2. Peripheral blood CD3 count > 200/µL by flow cytometry. Please note that this test might need to be repeated multiple times as standard practice to optimize collection efficiency.
3. Subjects will have a diagnosis of Diffuse Large B Cell Lymphoma (DLBCL), Follicular Lymphoma (FL), Mantle Cell Lymphoma (MCL), CLL, Marginal Zone Lymphoma (MZL), Lymphoplasmacytic Lymphoma (LPL) or B-ALL and will have failed at least 2 lines of therapy in the case of lymphoma and one line if the diagnosis is B-ALL or be refractory (no response or progressive disease) to first line therapy. A line of therapy must include conventional (immuno) chemotherapy (e.g. rituximab, cyclophosphamide, doxorubicin, and prednisone (R-CHOP) or Bendamustine plus Rituximab (BR) in the case of lymphoma) administered for at least 2 cycles. Second or greater lines of therapy must be administered for at least two cycles. Single agent anti-CD20 monoclonal antibody (e.g. rituximab, obinutuzumab) is not considered for the purposes of these criteria to count as a line of therapy. The definition of a line of therapy is taken according to recommended regimens for first and second line therapy in the relevant sections of the National Comprehensive Cancer Network (NCCN) guidelines. The most recent version of the guidelines will be used for eligibility determination. In the unlikely event that a subject received a first or second line regimen no longer listed in the most recent guidelines, but previously present in the version of the guidelines active at the time the therapy was administered, then the subject would be deemed to have received a line of therapy.
4. Subjects with pathological and clinical evidence of transformed indolent lymphoma (FL, CLL, MZL or LPL) are eligible for participation on this trial if they have received at least one line of therapy for transformed disease for at least two cycles regardless of response.
5. Demonstration of CD19 expression by immunohistochemistry or flow cytometry on a pathological specimen of lymphoma or ALL cells at any time in the course of prior treatment.
6. Subjects who are unable to receive commercially available CD19-CAR T-cell therapy.
7. Patients with lymphoma must have measurable or assessable disease. Patients in complete remission with no evidence of disease are not eligible.
8. Patients with B-ALL must have at least measurable detectable disease on two separate occasions at least 2 weeks apart to be eligible.
9. Subjects who relapse at > 100 days after autologous or allogeneic HSCT are eligible for participation on this trial. Allogeneic HSCT recipients must be off all immunosuppression for a minimum of 4 weeks before leukapheresis is performed and be free of active acute and chronic Graft Versus Host Disease (GVHD).
10. Subjects will be ≥ 18 and < 80 years of age.
11. Female subjects of childbearing potential must have a negative urine or serum pregnancy test and if sexually active must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive. Active contraception should continue for at least one year after CAR T-cell infusion.
12. Male participants must be willing to practice birth control from the time of enrollment on this study and for 6 months after receiving the preparative regimen.
13. Cardiac ejection fraction ≥ 0.45 by MUGA (multigated acquisition) or echocardiography.
14. No requirement for supplemental oxygen and no dyspnea at rest. DLCO (diffusing capacity of the lungs for carbon monoxide) and FEV (forced expiratory volume)1 ≥ 0.65 of predicted.
15. Karnofsky performance score ≥ 70.
16. Subjects must have an expected survival > 12 weeks.
17. Subjects must be able to comprehend the risks and methods used in this clinical trial and independently consent to participate.
18. Subjects must consent to anonymous reporting of data to the CIBMTR (Center for International Blood and Marrow Transplant Research).

Exclusion Criteria:

1. Infection with HIV (human immunodeficiency virus) and active viral replication. Patients with an undetectable viral load on ART (antiretroviral treatment) can be considered for participation on this protocol.
2. Infection with hepatitis B and active viral replication.
3. Infection with hepatitis C and active viral replication.
4. Active untreated CNS (central nervous system) leukemia or lymphoma. Patients with treated CNS leptomeningeal or parenchymal disease might be eligible if the CNS disease is inactive. The CSF (cerebrospinal fluid) must be clear on two separate occasions at least 4 weeks apart. Brain imaging must demonstrate no evidence of progressive disease on two separate occasions at least 4 weeks apart.
5. Active bacterial, fungal or viral infection.
6. Concurrent second malignancy requiring active therapy. Patients with breast or prostate cancer stable on hormonal therapy might be considered for participation if otherwise unimpaired.
7. Documented myocardial infarction within 6 months of study participation and/or symptomatic coronary artery or valvular disease or uncontrolled arrhythmia.
8. Investigational drug use within 30 days before leukapheresis.
9. Anti-cancer therapy administration within 4 weeks of leukapheresis including antiCD19 directed therapy, monoclonal antibody therapy, bi-specific T-cell engager therapy and targeted therapy such as Abelson tyrosine kinase inhibitors, Bruton's tyrosine kinase inhibitors, venetoclax and Lenalidomide or other IMiD (Immunomodulatory Drug).
10. Involved field radiation therapy is permitted if it terminates at least 15 days before leukapheresis and associated toxicity is grade 2 or less. Radiation therapy within 14 days of leukapheresis would make the subject ineligible.
11. Checkpoint inhibitor therapy within 4 weeks before leukapheresis.
12. Corticosteroid therapy at pharmacological dose (> 10 mg of prednisone or biological equivalent) within 4 weeks before leukapheresis.
13. Immunosuppressive therapy that cannot be stopped for 4 weeks prior to leukapheresis as deemed by the prescribing physician.
14. Laboratory abnormalities that indicate clinically significant hematological, hepatobiliary, or renal disease:

    AST (Aspartate transaminase)/SGOT(serum glutamic-oxaloacetic transaminase) > 2.0 times the upper limit of normal ALT (alanine aminotransferase)/SGPT (serum glutamic-pyruvic transaminase) > 2.0 times the upper limit of normal Total bilirubin > 2.0 times the upper limit of normal, unless subject has Gilbert's Syndrome (>3.0 times the upper limit of normal) Hemoglobin < 8 gm/dL or dependent upon transfusion to maintain ≥ 8 gm/dL White blood cell count < 2,000/mm3 Platelet count < 50,000/mm3 or dependent upon transfusion to maintain ≥ 50,000 mm Creatinine > 2.0 times the upper limit of normal or calculated creatinine clearance ≤ 40 mL/min.
15. Pregnant or lactating females.
16. Subjects who, in the opinion of the Investigator, will be non-compliant with study schedules or procedures.
17. Subjects who belong to a vulnerable population such as the homeless, the developmentally disabled and prisoners or have any condition that impairs their ability to provide informed consent or comply with study schedules or procedures.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2037-08-05 (Estimated); Study Completion 2037-12-01 (Estimated)

PRIMARY OUTCOMES:
Successful local CAR T-cell manufacturing | 48 months
  To demonstrate the feasibility of reliably producing CD19-targeted CAR T-cells at our site using the Prodigy device.
Safety of administration | 15 years
  To demonstrate the safety of administering the manufactured product to subjects as measured by adverse events.
Safety of administration | 30 days
  Cytokine Release Syndrome score
Safety of administration | 30 days
  Immune Effector Cell Associated Neurotoxicity Syndrome Grading for Adults (score) - A score of 10 represents no impairment, 7-9 grade 1 ICANS, 3-6 grade 2 ICANS, and 0-2 grade 3 ICANS. A score of 0 due to patient being unarousable and unable to perform assessment corresponds to grade 4 ICANS.
Safety of administration | 30 days
  Immune Effector Cell Associated Encephalopathy Score - A score of 10 represents no impairment, 7-9 grade 1 ICANS, 3-6 grade 2 ICANS, and 0-2 grade 3 ICANS. A score of 0 due to patient being unarousable and unable to perform assessment corresponds to grade 4 ICANS.

SECONDARY OUTCOMES:
Response to therapy | 48 months
  Response evaluation according to Lugano criteria for lymphoma and NCCN guidelines for ALL.
Response to therapy | 48 months
  Response criteria ALL-E and for MRD (minimal residual disease) ALL-F for B-ALL.
CAR T-cell kinetics | 100 days
  CAR T-cell counts by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: John Lister, MD, Principal Investigator — AHN
Locations (1):
- AHN Cancer Institute - West Penn Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No